CLINICAL TRIAL: NCT07327411
Title: A Single-arm, Multi-center, Prospective Clinical Study of Cetuximab β Combined With PRaG Regimen in the Treatment of EGFR-positive Advanced Refractory Solid Tumors
Brief Title: Cetuximab β Combined With PRaG Regimen in the Treatment of EGFR-positive Advanced Refractory Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK2025119-I01
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Advanced Refractory Solid Tumors
MeSH Terms: interventions — Radiation Dose Hypofractionation; Immune Checkpoint Inhibitors; envafolimab; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT+PD-L1+GM-CSF+EGFR (Experimental): Radiation: Hypofractionated radiotherapy 10-24Gy/5-8Gy/2-3f Drug1: PD-L1 inhibitor，Envafolimab 400mg，d1，q3w, until PD Drug2: GM-CSF 200μg, D1-D7,q3w, ≥8 cycles Drug3: anti-EGFR monoclonal antibody，cetuximab β 500mg/m2， d1， q3w, ≥8 cycles
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: PD-L1 inhibitor; Drug: GM-CSF; Drug: anti-EGFR monoclonal antibody

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 10-24Gy/5-8Gy/2-3f
Drug: PD-L1 inhibitor — 400mg，q3w, until PD
  Other Names: Envafolimab Injection
Drug: GM-CSF — 200μg, D1-D7, q3w，≥8 cycles
Drug: anti-EGFR monoclonal antibody — 500mg/m2 ，d1 ，q3w，≥8 cycles
  Other Names: cetuximab β

SUMMARY:
This study is a single-arm, multi-center, prospective clinical study aimed at exploring the efficacy and safety of cetuximab β combined with PRaG regimen in rescuing patients with EGFR-positive advanced refractory solid tumors.

DETAILED DESCRIPTION:
This study is a single-arm, multicenter, prospective clinical trial aimed at exploring whether adding cetuximab β to PRaG regimen is effective in patients with EGFR-positive, advanced, refractory solid tumors. The goal is to achieve efficient and durable tumor immune responses by precisely identifying tumor cells and overcoming tumor heterogeneity. By exploring new treatment models, the study seeks to open new avenues for the treatment of patients with advanced refractory solid tumors and improve patient outcomes. Patients who meet the inclusion and exclusion criteria will be treated according to the following protocol. Treatment will continue until disease progression or the occurrence of intolerable toxicity. Imaging assessments will be conducted every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign a written informed consent form;
* Age ≥18 years, male or female;
* Eligible patients must have recurrent or metastatic advanced solid malignancies, with a confirmed pathological diagnosis or medical history, and pathology showing EGFR positivity (IHC 1, 2, or 3; for colorectal cancer, RAS/BRAF wild-type patients can be enrolled if EGFR is negative), with no clear guideline-recommended standard treatment or intolerance to standard therapy, and with measurable metastatic lesions (>1 cm);
* Patient performance status is scored 0-3 according to the Eastern Cooperative Oncology Group (ECOG) criteria;
* Estimated life expectancy ≥3 months;
* No history of severe hematopoietic, cardiac, pulmonary, hepatic, or renal dysfunction or immunodeficiency;
* Good compliance.

Exclusion Criteria:

* Pregnant or breastfeeding women；
* Individuals with a history of other malignant diseases within the past 5 years, except for cured skin cancer and carcinoma in situ of the cervix；
* Individuals with uncontrolled epilepsy, central nervous system diseases, or psychiatric disorders, where the investigator judges that the clinical severity may hinder the signing of informed consent or affect patient compliance with medication；
* Clinically severe (i.e., active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure, or severe arrhythmias requiring medication, or a history of myocardial infarction within the past 12 months；
* Individuals requiring immunosuppressive therapy due to organ transplantation；
* Known significant active infection, or if the investigator judges there is a significant hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction, or other severe uncontrolled comorbid conditions；
* Individuals allergic to any component of the study drug；
* Individuals with a history of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, history of organ transplantation, or other immune-related diseases requiring long-term oral corticosteroid treatment；
* Individuals currently with acute or chronic tuberculosis infection (positive T-spot test, chest X-ray showing suspicious tuberculosis lesions)；
* Other situations deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate，ORR | Up to 2 years
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) u v1.1.

SECONDARY OUTCOMES:
progression free survival，PFS | Up to 2 years
  Time from cycle 1, day 1 of treatment to disease progression or death due to any cause
Disease control rate，DCR | Up to 2 years
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) o disease (SD) using RECIST v1.1.
Overall survival，OS | Up to 2 years
  Time from cycle 1, day 1 of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: liyuan zhang, PhD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No